CLINICAL TRIAL: NCT05157503
Title: "Epidemiology, Approaches to the Diagnosis and Treatment of Patients With Stage III Non-small Cell Lung Cancer in Russia"
Brief Title: Treatment of Patients With Stage III Non-small Cell Lung Cancer in Russia"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Autonomous Non-Profit Organization National Society of Onco-Pulmonologists (Other)
Responsible Party: Sponsor
Other Study IDs: 4
Record Dates: First submitted 2020-09-21; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Stage III Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In connection with the transition to the 8th version of the classification of lung cancer according to the TNM system, there are currently no precise epidemiological data on stage III NSCLC, clinical characteristics of patients in this group, approaches to therapy and treatment results in the Russian Federation. The published statistics only provide information on the overall incidence of stage III lung, trachea and bronchial cancer, which is about 40%. This observational study will make it possible to characterize the Russian population of stage III non-small cell lung cancer patients, approaches to choosing a treatment option for stage III NSCLC and the outcomes of this treatment in real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- stage III non-small cell lung cancer

Exclusion Criteria:

- the rest of the disease stage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with morphologically proven stage III non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Examine clinical and morphological groups | 10/01/2023
  * gender ratio (husband, wife)
  * smoking status (smoker, non-smoker, past smoker)
  * proportional distribution: squamous cell, adenocarcinoma, dimorphic cancer, others)
  * how many patients with mediastinal lymph node involvement: (N0, N1, N2, N3)
  * detection frequency: PDL (PDL <1, PDL> 1, PDL <49, PDL> 50), EGFR (EGFR + (19.24 exon) EGFR-), (ALK +, ALK -), (ROS-1 +, ROS-1 -) Get information about regional algorithms
  * Variants of treatment tactics:
  Percentage:
  a. Surgery
  v. Chemotherapy
  -Diagnostic algorithm:
  a. Morphological verification frequency b. The frequency of confirmation of metastatic lesions within the thoracic lymph nodes c. F

SECONDARY OUTCOMES:
Explore clinical approaches | 10/01/2023
  * Percentage of treatment options depending on:
    a. histological type
  * squamous
  * adenocarcinoma
  * dimorphic
  * 3 A st
  * 3B st
Diagnostic algorithm: | 10/01/2023
  v. from a variant of molecular genetic disorders
  * PDL <1
  * PDL> 1
  * PDL <49
  * PDL> 50
  * EGFR +
Percentage of treatment options | 10/01/2023
  from functional status
  * ECOG 1
    1. only surgical treatment
    2. surgical + drug treatment
    3. surgical + drug treatment + radiation therapy
    4. drug treatment
    5. drug treatment + radiation therapy
    6. radiation therapy
  * ECOG 2
    1. only surgical treatment
    2. surgical + drug treatment
    3. surgical + drug treatment + radiation therapy
    4. drug treatment
    5. drug treatment + radiation therapy
    6. radiation therapy
  * ECOG 3
    1. only surgical treatment
    2. surgical + drug treatment
    3. surgical + drug treatment + radiation therapy
    4. drug treatment
    5. drug treatment + radiation therapy
    6. radiation therapy

OTHER OUTCOMES:
-Evaluate the frequency of decision-making as a standard practice vs with an individual decision | 10/01/2023
  * Percentage of treatment options depending on:
    a. The nature of the progression
  * oligo progression
  * systemic progression
    b. Prior treatment options v. after surgical treatment
    d. Afte

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center of Oncology. N. N. Blokhin, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided